CLINICAL TRIAL: NCT01544036
Title: Monitoring Renal Blood Flow Using Contrast Enhanced Ultrasound in Predicting Acute Kidney Injury After Exposure to Iodinated Contrast Agent
Brief Title: Monitoring Renal Blood Flow With Contrast Enhanced Ultrasound During Coronary Angiogram
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15591; K23DK074616 (NIH)
Record Dates: First submitted 2012-02-27; First posted 2012-03-05 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Contrast Induced Acute Kidney Injury
Keywords: AKI; contrast nephropathy; renal blood flow
MeSH Terms: interventions — perflutren

ARMS (1):
- Contrast Enhanced Ultrasound (Experimental): Renal blood flow before and after exposure to iodinated contrast agent (perflutren) also known as Definity will be measured using contrast enhanced ultrasound (CEUS).
  Interventions: Drug: perflutren

INTERVENTIONS:
Drug: perflutren — Contrast Enhanced Ultrasound is performed during continuous intravenous infusion of Definity (drug) to assess changes in renal blood flow during the study
  Other Names: Definity

SUMMARY:
Contrast induced nephropathy (CN) is a common cause of acute kidney injury and is associated with increased morbidity and mortality and healthcare cost. Iodinated contrast media (ICM) induce kidney injury through vasoconstriction and ischemia as well as direct tubular toxicity. Older subjects, individuals with preexisting kidney disease, diabetes, hypotension, and those exposed to higher volumes of ICM are at higher risks for CN. Within the last several years, multiple strategies have been used in clinical studies to reduce the risk of CN in high risk individuals with inconsistent results. In general, it is agreed that volume expansion is effective in reducing the risk. However, no study has looked at changes in renal blood flow (RBF) in response to volume expansion or after exposure to ICM to investigate its relationship with occurrence of CN.

In this proposal, up to 125 individuals with preexisting kidney disease as evidenced by an estimated glomerular filtration rate (eGFR) between 30 - 60 ml/min/1.73 m2 and up to 25 individuals with normal renal function (total of up to 150 individuals) who are scheduled for coronary angiography will be studied. Each individual will have serial measurements of RBF; at baseline, after volume expansion with normal saline, and after exposure to ICM, using the novel technique of contrast enhanced ultrasound (CEU). The investigators will investigate the utility of monitoring RBF with CEU in predicting the occurrence of CN (a rise of > 0.3 mg/dL or 25% in baseline serum creatinine 48 hours after exposure to ICM) after adjusting for other known risk factors in the group of subjects with reduced GFR. The investigators will also examine the correlation between RBF changes and other urinary and serum biomarkers of kidney injury in this group. Up to 25 individuals with a normal kidney function will be studied in a separate part of the study in which the accuracy of CEU based measurements of RBF will be compared to the RBF and blood flow velocity obtained simultaneously using a Doppler flow probe placed directly inside the main renal artery during coronary angiogram procedure. Total to enroll = 150.

DETAILED DESCRIPTION:
What will be done in this protocol? Specific to Aim 1: To investigate the correlation between changes in RBF after exposure to iodinated contrast agent, measured by CEU, on occurrence of acute kidney injury (AKI) in a population of subjects at risk for CN.

Procedures: Subjects with an estimated glomerular filtration rate (eGFR), measured by the Modification of Diet in Renal Disease (MDRD) formula, between 30 - 60 ml/min/1.73 m2 who are scheduled for a coronary angiogram will be enrolled in this study. These subjects are considered to be at higher risks of CN. It is important to clarify that all subjects are scheduled for a coronary angiography for clinical reasons before enrollment in this study. Coronary angiography is not a part of interventions of this protocol. The decision regarding the need for coronary angiography and the strategies for its prevention are made by the subjects' healthcare providers and not the research team.

The details of protocol will be discussed with all interventional cardiologists and permission will be obtained to discuss study details with potential subjects. Eligible subjects will be identified by searching the electronic medical record of individuals who are listed in the cardiac catheterization laboratory schedule for inclusion and exclusion criteria. Subjects who appear to qualify for study participation based on medical record review the inclusion and exclusion criteria will be approached. The details of the study goals, procedures and risks will be discussed with each individual and questions will be answered. The subjects will then be asked to sign the informed consent form. They will then be enrolled in the study.

Since undergoing an X-ray examination or exposure to iodinated contrast media are contraindicated in pregnancy, we assume all women of child bearing age having a test to rule out pregnancy before enrolling in the study. If this test is not done, we will contact the subject's cardiologist and arrange for it as a part of clinical care and not a research related procedure.

At the time of enrollment data on subjects' age, race, gender, ethnicity, history of coronary artery disease, diabetes and congestive heart failure will be collected. Subjects with a history of heart failure will be asked about presence of symptoms of heart failure such as shortness of breath at rest or with activities, fatigue, palpitation and dyspnea. This information will be used to identify the New York Heart Association (NYHA) class of heart failure which is considered a risk factor for CN. List of medications used by subjects will also be recorded. Vital signs will be recorded.

Blood samples for basic metabolic panel and urine samples for urinalysis will be collected and sent to the University of Virginia lab. More blood and urine samples will be collected for measurement of the concentrations of biomarkers of kidney injury neutrophil gelatinase-associated lipocalin (NGAL), cystatin C, beta 2 microglobulin, epithelial growth factor (EGF), uromodulin, osteopontin, albumin and creatinine. These samples will be sent to the the O'Brien Center at the University of San Diego, California for analysis..

Baseline 2-dimensional kidney ultrasound images will be obtained. All study subjects will undergo baseline contrast enhanced ultrasound imaging of the kidneys using Definity intravenous infusion as described in details below. They will then receive intravenous infusion of normal saline for prevention of CN. Please see "hydration protocol" below.

Immediately before transfer to the cardiac catheterization lab and after volume expansion with i.v. normal saline, CEU imaging of the kidneys using Definity will be repeated.

Subjects will undergo coronary angiogram procedure as planned by their interventional cardiologists. Immediately after this procedure, CEU imaging of the kidneys using Definity will be repeated. Subjects will be monitored for a minimum of 30 minutes after completion of Definity infusion. Blood samples for basic metabolic panel and urine samples for urinalysis will be collected and sent to the UVA lab. The research study procedures for this visit will end at this time. Routine cardiac catheterization lab procedures will be followed at this time.

Information on the volume and type of ICM will be recorded. Subjects will be discharged as scheduled by the cardiology team. One to three days (24 - 72 hours) later the subjects will return for a follow up visit. During the follow up visit, questions will be asked to assess for potential adverse events. Vital signs will be obtained (blood pressure and heart rate). Blood samples for basic metabolic panel and urine samples for urinalysis will be collected and sent to the UVA lab. More blood and urine samples will be collected for measurement of the concentrations of biomarkers of kidney injury NGAL, cystatin C, beta 2 microglobulin, EGF, uromodulin, osteopontin, albumin and creatinine. These samples will be sent to the O'Brien Center at the University of San Diego in California.

The outcome of the study, AKI, will be defined as a rise of greater than 0.3 mg/dL or 25% in the baseline serum creatinine concentration 48 hours after exposure to ICM.

Specific Aim 2: To validate the RBF data obtained by CEU by comparing it to measurements obtained by a Doppler ultrasound probe placed inside the main renal artery.

Procedures: Up to 25 subjects with normal renal functions who are scheduled for a coronary angiography will be studied in this part of the proposed study. Blood samples for basic metabolic panel and urine samples for urinalysis will be collected and sent to the UVA lab.

Immediately before undergoing coronary angiography, each subject will undergo CEU study using Definity to measure baseline RBF. Femoral or radial access has already been obtained to perform the coronary angiogram. A guide catheter is used to selectively engage the renal artery and 5 cc of contrast will be injected to perform renal angiography. If the renal artery appears angiographically normal and is without evidence of any degree of atherosclerotic renal artery stenosis, then a Doppler flow wire (0.014") will be advanced into the main renal artery. If the patient is not already systemically anticoagulated for the coronary angiogram or coronary intervention, then heparin is administered (50 U/kg) to prevent clotting on the Doppler wire. Proper positioning of the Doppler wire will be confirmed by injecting 1-2 cc of contrast. Velocity of the blood flow within the main renal artery will be measured directly using this Doppler wire. After completion of these measurements, coronary angiography procedures will be performed as scheduled. Measurement of blood velocity in the main renal artery with the Doppler probe will be repeated before removal of the arterial catheter. CEU using Definity for measurement of RBF will be repeated at this point. Subjects will be monitored for a minimum of 30 minutes after completion of Definity infusion and a urine sample will be obtained and sent to the UVA lab for urinalysis. Blood samples for basic metabolic panel will be collected and sent to the UVA lab. The changes from baseline in the velocity of blood after exposure to ICM obtained by Doppler probe will be compared to the values obtained by CEU. Multiple measurements (at least three) using each method will be performed at each time point and the mean of these measurements will be compared.

Contrast Enhanced Ultrasound Subjects will be connected to a continuous pulse oximeter and heart monitor. The Definity vial will be placed at room temperature before being used. It will be activated after shaking the vial using Vialmix for 45 seconds. It will be used immediately after activation. 1.3 mL of Definity will be mixed in 30 ml of preservative free saline. Infusion of Definity into a peripheral vein will be started at 2 ml/min and titrated for optimal image quality (not to exceed 10 ml/min at any time). After reaching steady state (2 -3 minutes) baseline contrast ultrasound imaging of right kidney will be performed with low mechanical index (MI) of 0.1. High MI (1.0) impulse will be used to disrupt Definity microbubbles within the kidney tissue. This would result in a very brief time period during which renal cortex is free of microbubbles and appears completely anechoic (time zero). As continuous infusion of microbubbles continues, during the wash-in period renal tissue is replenished with microbubbles. Time-intensity curve after disruption of tissue microbubbles will be fitted to a rising exponential function: intensity (y) = basic intensity (BI) + A [1-exp(-beta.t) using specialized software. The slope of this curve or beta is related to the velocity of microbubbles (or blood) that enter the tissue and the plateau of the curve or A is related to the relative blood volume within the tissue. Since blood flow is the movement of a certain volume of blood at a certain speed, the product of the two (A.beta) would represent tissue blood flow. After disruption of microbubbles within the kidney tissue with a high MI pulse, continuous imaging of the kidney with low MI (0.1) will continue for about 15- 30 seconds to generate the time-intensity graph. The high MI pulse and replenishment sequence will be repeated two more times. An average of the three parameters obtained at each time period will be used for the final analysis. Infusion of Definity will stop at this point. A urine sample will be collected for urinalysis after 30 minutes of stopping Definity to assess for potential renal related adverse events.

Hydration Protocol:

0.9% sodium chloride (normal saline) solution will be infused intravenously at a rate of 3 mL/kg/hr for one hour. This will be followed by normal saline given at a rate of 1 ml/kg/hr for the remainder of the time before and also during and at least for one hour after coronary angiogram. Patients with heart failure and documented ejection fraction of < 30% will receive normal saline infusion at a reduced rate of 1.5 ml/kg/hr for the 1st hour followed by 0.5 mL/kg/hr after that for the same time periods as for other subjects. At any point, if a subject experiences shortness of breath, oxygen saturation will be measured and intravenous hydration protocol will be stopped.

ELIGIBILITY:
Inclusion For specific aim 1 - Subjects with reduced kidney function

1. Adult (>18 years of age) men and women
2. All races and ethnicities
3. Chronic kidney disease stage 3 with an estimated GFR by MDRD formula between 30 - 59 ml/min/1.73 m2
4. Being scheduled for a coronary angiography study as part of their clinical care

For specific aim 2 - Subjects with normal kidney function

1. Adult (>18 years of age) men and women
2. All races and ethnicities
3. Being scheduled for a coronary angiography study
4. Estimated GFR greater than or equal to 60 ml/min/1.73 m2

Exclusion For specific aim 1 - Subjects with reduced kidney function

1. Estimated GFR greater than 60 or below 30 ml/min/1.73 m2
2. History of kidney transplantation
3. Known history of a right to left intracardiac shunt
4. Pregnancy or lactation
5. History of allergies to Definity®
6. History of Pulmonary Hypertension

For specific aim 2 - Subjects with normal kidney function

1. Estimated GFR less than 60 ml/min/1.73 m2
2. History of kidney transplantation
3. History of a right to left intracardiac shunt
4. Pregnancy or lactation
5. History of allergies to Definity®
6. History of recent major bleeding
7. History of allergy to heparin or heparin-induced thrombocytopenia
8. History of renal artery stenosis
9. Evidence of renal artery stenosis during the placement of Doppler wire in the renal artery
10. History of Pulmonary Hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | 24 - 72 hours
  Correlation between changes in renal blood flow measured by contrast ultrasound and occurrence of AKI.

SECONDARY OUTCOMES:
Change in novel biomarkers of AKI | 24 - 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States